CLINICAL TRIAL: NCT00000836
Title: A Phase II/III Trial of Human Anti-CMV Monoclonal Antibody MSL 109 (MACRT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Purpose: Treatment
Other Study IDs: ACTG 294
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-10

CONDITIONS: Cytomegalovirus Retinitis; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome; Antibodies, Monoclonal; Cytomegalovirus Retinitis
MeSH Terms: conditions — Cytomegalovirus Retinitis; HIV Infections; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome | interventions — sevirumab

INTERVENTIONS:
Drug: Sevirumab

SUMMARY:
To compare the safety and efficacy of sevirumab (MSL 109; Protovir), human anti-cytomegalovirus (CMV) monoclonal antibody, plus active primary treatment versus placebo plus active primary treatment in AIDS patients with newly diagnosed and relapsed CMV retinitis.

Ganciclovir and foscarnet are used for treatment of CMV retinitis, but cause hematologic toxicity and nephrotoxicity, respectively. Despite continued maintenance therapy with these drugs, relapse occurs in 85 percent of patients within 4 months. Studies suggest that MSL 109, a human monoclonal antibody, when given with either ganciclovir or foscarnet, may increase initial response and prolong time to progression in patients with CMV retinitis.

DETAILED DESCRIPTION:
Ganciclovir and foscarnet are used for treatment of CMV retinitis, but cause hematologic toxicity and nephrotoxicity, respectively. Despite continued maintenance therapy with these drugs, relapse occurs in 85 percent of patients within 4 months. Studies suggest that MSL 109, a human monoclonal antibody, when given with either ganciclovir or foscarnet, may increase initial response and prolong time to progression in patients with CMV retinitis.

Patients are randomized to receive either MSL 109 or placebo every 2 weeks as supplemental therapy to primary CMV treatment.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication: Required:

* Primary CMV treatment.

Patients must have:

* AIDS.
* Active CMV retinitis.
* At least one photographable lesion of one-quarter or more optic disc area in size.
* Undergoing primary treatment for CMV retinitis that is not contraindicated with MSL 109.
* Visual acuity in at least one eye of 3 or more letters on Early Treatment Diabetic Retinopathy Study ( ETDRS ) chart at 1 meter distance ( Snellen equivalent 5/200 ). Note:
* Exceptions may be made if visual acuity impairment is possibly reversible and there is at least light perception in that eye.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Retinal detachment not scheduled for surgical repair.
* Media opacity that precludes visualization of the fundus.
* Active medical problems sufficient to hinder study compliance.

Concurrent Medication:

Excluded:

* IVIG.
* CMV immune globulin ( CMVIG ).
* Interferon alpha.
* Interferon gamma.
* Interleukin-2 ( IL-2 ).

Drug or alcohol abuse sufficient to hinder study compliance.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300
Dates: Study Completion 1998-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - UCSD - Shiley Eye Ctr / SOCA, La Jolla, California
  - UCLA - Jules Stein Eye Institute / SOCA, Los Angeles, California
  - UCSF - San Francisco Gen Hosp, San Francisco, California
  - Northwestern Univ / SOCA, Chicago, Illinois
  - Johns Hopkins Hosp / SOCA, Baltimore, Maryland
  - New York Univ Med Ctr / SOCA, New York, New York